CLINICAL TRIAL: NCT04274946
Title: The Comparative Analysis of Multimodal Markers to Identify Sentinel Lymph Node in Breast Cancer
Brief Title: Sentinel Lymph Node Biopsy With Hybrid Technique in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Guldeniz Karadeniz Cakmak, Head of General Surgery Departmet, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-09-09
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: breast; sentinel lymph node; patent blue; indocyanine green
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RAI+PB+US (Active Comparator): Sentinel lymph node mapping with dual tracer (radioisotope and patent blue) and intraoperative ultrasound to identify SLN in the breast cancer patients
  Interventions: Procedure: Sentinel lymph node biopsy
- RAI+ICG+US (Experimental): Sentinel lymph node mapping with dual tracer (radioisotope and ICG) and intraoperative ultrasound to identify SLN in the breast cancer patients
  Interventions: Procedure: Sentinel lymph node biopsy
- RAI+PB+ICG+US (Experimental): Sentinel lymph node mapping with triple tracer (radioisotope,ICG and patent blue) and intraoperative ultrasound to identify SLN in the breast cancer patients
  Interventions: Procedure: Sentinel lymph node biopsy
- PB+ICG+US (Experimental): Sentinel lymph node mapping with triple tracer (ICG and patent blue) and intraoperative ultrasound to identify SLN in the breast cancer patients
  Interventions: Procedure: Sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy — Sentinel lymph node biopsy(SLNB) procedure with different mapping methods using combination of radioactive colloid, patent blue, indocyanine green associated with intraoperative ultrasound.

SUMMARY:
Sentinel lymph node (SLN) biopsy is the gold standard method to stage axilla in breast cancer. The aim of the study is to compare the efficiency of various methods to identify SLN is breast cancer patients.

DETAILED DESCRIPTION:
Various markers has been used for SLN biopsy including isosulfan blue (patent blue), indocyanine green (ICG), radioisotope colloid (RAIC) and ultrasound (US) with several advantages and disadvantages. In this study investigators designed an algorithm using the combination of mapping with patent blue, ICG, RAIC and US to compare the accurate identification of SLN in breast cancer patients. The protocol is based on the hypothesis that identification rate of SLN is increased with multiple agents. Patent blue and ICG provides visual guidance. The combination of dyes with sonographic and RAIC method have the potential to prevent obstacles and ensure better outcomes as an identification strategy.

Patent blue provides visual identification of the SLN. ICG fluorescence can be detected percutaneously and by means of fluorescence imaging system in real time. RAI has several advantages, but disadvantages as well, like cost and invisibility. RAI can only be detected and confirmed by means of sound and numerical value through gamma probe. All breast cancer patients underwent axillary ultrasound before SLNB with different mapping combinations. The determination of abnormal axillary lymph node was followed by ultrasound-guided FNA cytology of these nodes. The sonographic abnormality criteria of the nodes were defined as; completely hypoechoic node, asymmetric focal hypoechoic node, cortical lobulation more than 3, cortical thickness >2mm, totally spheric appearance, absence of fatty hilum and compromise of normal vascularity (hypervascularization from various poles). Patients with negative results of FNA would undergo SLNB. Lymphatic mapping was performed with abovementioned dyes and radioactive colloid. Before the incising for SLNB real time intraoperative US was performed and suspicious axillary lymph nodes were seen by ultrasound guidance. In the SLNB operation, radioactive or dyed nodes and sonographically suspicious nodes were removed and labeled separately for pathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary breast cancer by core needle, incisional or excisional biopsy
* cN0 patients
* In patients with abnormal axillary lymph nodes sonographically US-guided FNA cytology of these nodes were performed and FNA cytology negative patients planed to undergo SLNB with different mapping techniques.

Exclusion Criteria:

* Patients with neoadjuvant therapy
* Patients with pathological diagnosed ductal carcinoma in situ by excisional biopsy
* Patients with pathologically proven axillary disease
* Patients with T4d tumor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Identification rate of sentinel lymph node | During operation
  The ability to identify a sentinel lymph node successfully with different mapping techniques

SECONDARY OUTCOMES:
Average number of excised sentinel lymph nodes | Histological report expected within an average of 2 weeks after sentinel lymph node biopsy
  The effect of mapping technique on the number of excised nodes
False-negative rate of axillary US | Histological report expected within an average of 2 weeks after sentinel lymph node biopsy
  False negative rate for SLN surgery in women with normal or axillary US and at least 2 SLNs were excised, defined as the number of patients with no positive lymph nodes by SLN and with at least one positive lymph node by axillary lymph node dissection divided by the total number of patients with at least one positive lymph node by SLN or ALND multiplied by 100, or vise versa. For abnormal axillary US, false negative rate is calculated similarly.
Morbidity | 36 months
  Lymphedema, shoulder movement pain, or functional deformity after SLNB with different mapping techniques will be assessed by clinicians during follow-up with 3 months periods. The result will be the percentage of patients which suffer from some complications after SLNB or AD. Common morbidity rate after AD is 20%, after SLNB 1-2%.

CONTACTS AND LOCATIONS:
Overall Officials: Güldeniz Karadeniz Cakmak, MD, Study Chair — Bülent Ecevit University Department of Surgery; Rabiye Uslu Erdemir, MD, Study Director — Bülent Ecevit University Department of Nucleer Medicine; Hakan Bakkal, MD, Principal Investigator — Bülent Ecevit University Department of Radiation Oncology; Hüseyin Engin, MD, Principal Investigator — Bülent Ecevit University Department of Clinical Oncology
Locations (1):
- Bülent Ecevit University, Zonguldak, Turkey (Türkiye)